CLINICAL TRIAL: NCT02082483
Title: Pilot Study to Determine Feasibility of a Randomized Trial of Screening for Coronary Artery Disease in Kidney Transplant Candidates
Brief Title: Coronary Artery Disease Screening in Kidney Transplant Candidates
Acronym: CADScreening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Gill, Dr. John Gill, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-00141; MOP 133509 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease; Coronary Artery Disease
Keywords: Kidney Transplant; Screening
MeSH Terms: conditions — Kidney Failure, Chronic; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective Screening (Experimental): Patients randomized to selective-use of screening tests will not routinely undergo Myocardial Perfusion Scintography or Dobutamine Stress Echocardiography. If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.
  Interventions: Other: Selective Screening
- Regular Screening (No Intervention): Patients randomized to regular screening will be tested as per the current standard described in guidelines published by the National Kidney Foundation (e.g. annually while wait-listed for transplantation). If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.

INTERVENTIONS:
Other: Selective Screening — Patients randomized to selective-use of screening tests will not routinely undergo Myocardial Perfusion Scintography or Dobutamine Stress Echocardiography. If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.
  Arms: Selective Screening

SUMMARY:
Kidney transplant candidates are at very high risk for coronary artery disease (CAD). The optimal strategy to monitor and maintain the cardiac fitness of patients awaiting kidney transplantation is unknown. Currently patients undergo annual testing; however, screening for CAD may increase morbidity and mortality by:

1. exposing patients to the risk of angiography and revascularization procedures
2. delaying or excluding patients from life saving transplantation.

Before proceeding with a definitive study to determine whether screening is necessary, feasibility will be determined in this pilot study.

DETAILED DESCRIPTION:
This pilot trial will determine the feasibility of a multi-center, randomized, parallel group definitive trial. Asymptomatic wait-listed patients will be randomized to routine screening for coronary artery disease (CAD) (i.e. Myocardial Perfusion Scintigraphy (MPS) or Dobutamine Stress Echo (DSE)) as per the current standard of care versus selective screening based on symptoms. Patients enrolled in the pilot will be included in the definitive trial analysis. The pilot trial will include four Canadian centres. The definitive trial will aim to determine if a strategy of selective use of screening tests (i.e. Myocardial Perfusion Scintigraphy or Dobutamine Stress Echo) only in the presence of symptoms (i.e. chest pain, dyspnea etc) is non-inferior with respect to the composite endpoint of non-fatal MI and cardiac death compared to screening all asymptomatic wait-listed patients at regular intervals as described in transplant specific guidelines published by the National Kidney Foundation.

Currently there is no strong evidence for or against using routine cardiac screening of asymptomatic transplant patients, more evidence based randomized clinical trials are needed. This need is further highlighted by a number of factors such as: wait-listed patients are increasing in number and medical complexity; longer wait times and changing donor characteristics can increase CAD risk; wait-listed patients are at high risk for CAD but are commonly asymptomatic; the standard of care is not evidence based and is expensive; the current standard may be harmful. The study will determine feasibility of a definitive trial through the measures outlined under 'Outcome Measures'.

End stage renal disease (ESRD) patients wait-listed for kidney transplantation will be randomized to undergo selective screening for CAD, in which patients are only screened if they develop symptoms suggestive of CAD or the current standard of care that involves regular screening for CAD at fixed time intervals based on the presence of risk factors. Patients will remain on the pilot trial protocol until death, non-fatal MI, transplantation, permanent removal from the waiting list for any reason, or 24 months after enrolment in the pilot trial. During wait-listing, follow-up telephone interviews and chart reviews will be performed every six months. After transplantation, an in-person follow up visit and chart review will occur at the time of discharge from hospital, and a telephone interview and chart review will be performed 3 months after transplantation. Patients will be followed for 24 months from the date of enrolment. Patients who receive a kidney transplant during the study will be followed for 27 months.

For the pilot trial, descriptive analyses are planned. Feasibility will be summarized with proportions, rates, means, and medians as appropriate. Comparison of the definitive trial outcomes between treatment groups, will not be done at the end of the internal pilot as these patients will be included in the definitive trial. Analyses of enrolment rates and consent rates will be done after the enrolment phase of the pilot trial in late 2014. An interim analysis of protocol adherence is planned in mid 2016 in support of the definitive trial funding application in September, 2016.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* active on the deceased donor transplant waiting list

Exclusion Criteria:

* patients not expected to require further screening for CAD prior to transplantation by the current standard of care. For example, a diabetic patient recently screened for CAD and expected to be transplanted <12 months from the start of the study would not require further screening according to current guidelines and would be ineligible
* patients with signs or symptoms suggestive of active cardiac disease such as unstable coronary syndromes, de-compensated heart failure, uncontrolled arrhythmia, and severe valvular heart disease
* patient who have been put "on hold" for transplantation due to a medical problem (e.g. an infection)
* prior extra-renal transplant recipients
* multi-organ transplant candidates (e.g. kidney pancreas transplant candidates)
* patients with a planned living donor transplant
* patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gill, MD, Principal Investigator — St. Paul's Hospital
Locations (6):
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Selective Screening | Regular Screening
Started | 71 | 73
Completed | 65 | 67
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selective Screening | Regular Screening | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.80 [45.31 to 63.38] | 54.98 [46.33 to 60.68] | 52.26 [42.79 to 61.84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 33 | 56
  Male | 48 | 40 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Aboriginal | 1 | 1 | 2
  Asian | 14 | 8 | 22
  Black | 8 | 2 | 10
  Caucasian/White | 29 | 18 | 47
  Indian Sub-continent | 6 | 1 | 7
  Mid East/Arabian | 4 | 3 | 7
  Pacific Islander | 4 | 3 | 7
  Unknown | 2 | 2 | 4
  Other/Multiracial | 3 | 3 | 6
Cause of End-Stage Renal Disease (ESRD) [Count of Participants; unit: Participants]
  Diabetes Mellutis | 15 | 18 | 33
  Polycystic Kidney Disease | 8 | 9 | 17
  Glomerulonephritis | 23 | 20 | 43
  Hypertension | 2 | 4 | 6
  Other/Unknown | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Adhering to the Expected Number of Screening Tests
Description: Adherence will be defined by completion of the expected number of screening tests during follow up as per the 2005 National Kidney Foundation guidelines. For example, the expected number of screening tests in a diabetic patient who did not develop symptoms would be zero in the selective screening group, while the same patient would be expected to completed two screening tests if randomized to regular screening. Tests performed for clinical symptoms of CAD will be excluded from the determination of adherence.
Time Frame: Up to 27 months
Measure: Number; unit: participants
Arm/Group | Selective Screening | Regular Screening
Number analyzed (Participants) | 71 | 73
participants | 59 | 71

2. Primary Outcome: Enrolment Rates
Description: The total number of subjects enrolled across all sites will be monitored monthly from the CRO, Ottawa Hospital Research Institute (OHRI), which issues the randomization scheme.
Time Frame: Measured after enrolment period of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Selective Screening | Regular Screening
Number analyzed (Participants) | 71 | 73
Participants
  St. Paul's Hospital | 15 | 16
  Vancouver General Hospital | 12 | 12
  Ottawa Hospital Research Institute | 21 | 21
  McGill | 7 | 9
  University Health Network | 10 | 8
  St. Joseph's Health Centre | 6 | 7

3. Primary Outcome: Consent Rate
Description: The percentage of patients willing to participate will be established at each site. Willingness to enrol in the study will be recorded on each patient's case report form along with the reason for any refusal to consent.
Time Frame: Measured after enrolment period of 6 months
Population: Number of participants approached to consent to study.
Measure: Count of Participants; unit: Participants
Groups:
- Selective or Regular Screening: Patients to be randomized to selective-use of screening tests will not routinely undergo Myocardial Perfusion Scintography or Dobutamine Stress Echocardiography. If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.
  Selective Screening: Patients randomized to selective-use of screening tests will not routinely undergo Myocardial Perfusion Scintography or Dobutamine Stress Echocardiography. If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.
  Patients randomized to regular screening will be tested as per the current standard described in guidelines published by the National Kidney Foundation (e.g. annually while wait-listed for transplantation). If patients develop symptoms of CAD at any time, they will undergo investigations as per the usual standard of care.
Arm/Group | Selective or Regular Screening
Number analyzed (Participants) | 211
Participants
  Consented | 144
  Declined | 67

4. Secondary Outcome: Number of Participants With Cardiac Events
Description: A composite outcome of cardiac death and non-fatal myocardial infarction will be looked at and adjudicated by a blinded clinical endpoints committee.
Time Frame: Up to 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Selective Screening | Regular Screening
Number analyzed (Participants) | 71 | 73
Participants
  Cardiac Death | 0 | 0
  Non-Fatal Myocardial Infarction | 4 | 3

5. Other Pre Specified Outcome: Number of Participants With Transplant Events
Description: Patient transplantation will be documented on the subject case report form.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Selective Screening | Regular Screening
Number analyzed (Participants) | 71 | 73
Participants | 36 | 39

6. Other Pre Specified Outcome: Number of Participants With Wait List Holds or Removals
Description: Indication for hold or removal will be measured as well.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Selective Screening | Regular Screening
Number analyzed (Participants) | 26 | 24
Participants
  Wait List Holds | 22 | 20
  Wait List Removals | 4 | 4

7. Other Pre Specified Outcome: Number of Health Care Encounters
Description: The information captured will include outpatient, day care, and emergency room use (including any diagnostic testing and all medical and surgical interventions (i.e. use of thrombolytics, revascularization procedures), inpatient encounters and resource utilization (hospitalizations, procedural costs), physician consultations. Indirect patients costs (time off work, transportation costs), and quality of life (measured using the short-form 36 (SF36).
Time Frame: Up to 27 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected 24 months from the date of enrollment and 3 months after transplantation date for those patients transplanted.
Description: During each follow up visit, participants were reviewed/asked if any of the following adverse events happened: death, myocardial infarction, non-fatal cardiac arrest, stroke, bleeding, coronary angiogram, revascularization, and hospitalization ≥ 24 hours.
Arm/Group | Selective Screening | Regular Screening
All-Cause Mortality (participants affected / at risk) | 2/71 | 3/73
Serious Adverse Events (participants affected / at risk) | 20/71 | 18/73
Other Adverse Events (participants affected / at risk) | 22/71 | 17/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selective Screening (N=71) | Regular Screening (N=73)
Bleeding (Blood and lymphatic system disorders) | 3 | 6
Coronary Angiogram (Cardiac disorders) | 5 | 3
Death (Investigations) | 2 | 3
Non-Fatal Cardiac Arrest (Cardiac disorders) | 3 | 1
Myocardial Infarction (Cardiac disorders) | 4 | 3
Revascularization (Vascular disorders) | 3 | 1
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selective Screening (N=71) | Regular Screening (N=73)
Non-Transplant Hospitalization (Investigations) | 22 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02082483/Prot_SAP_000.pdf